CLINICAL TRIAL: NCT04630938
Title: Effects of Anesthetics on Inflammatory Markers in Patients Undergoing Abdominal Surgeries.
Brief Title: Effects of Anaesthesia on Inflammatory Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esam Hamed, clinical professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17300478
Record Dates: First submitted 2020-07-12; First posted 2020-11-16 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Inflammatory Response
MeSH Terms: interventions — Morphine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G-M (Active Comparator): Received classic general Anesthesia, intrathecal (Bupivacaine 15 mg, morphine 4 microgram/kg) plus saline infusion intraoperative and postoperative.
  Interventions: Drug: Morphine Sulfate
- G-ML (Active Comparator): Received classic general Anesthesia, intrathecal morphine in a dose of 4 microgram/kg, and intravenous lidocaine in a loading dose of 1.5 mg/kg, then 2 mg/min with the saline infusion over the time of the operation and the next 4 hours postoperative.
  Interventions: Drug: morphine+lidocaine
- G-0 (Placebo Comparator): Received General Anesthesia and Spinal anesthesia as previously described with saline infusion in the same design as in the previous two groups.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Morphine Sulfate — intrathecal morphine will be added to anaesthetics
  Arms: G-M
Drug: morphine+lidocaine — local anesthetic will be infused intravenously
  Arms: G-ML
Drug: Saline — intravenous saline infusion
  Arms: G-0

SUMMARY:
undertake confidently both open and laparoscopic cholecystectomy. Major types of body injuries surgical or accidental; evoke a temporary, yet predictable systemic inflammatory response caused by hormonal, immunological and metabolic mediators. This inflammatory response is essential for tissue repair and has evolved to maximize the organisms' healing potential. In healthy individuals the inflammatory response to major surgery is well balanced consisting of pro- and anti-inflammatory mediators. The severity of injury, the occurrence of surgical complications and its accompanying level of stress may hinder the balance of the inflammatory response6.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aging 18 - 55 years old
* Patients scheduled for abdominal surgeries
* Patients with American Society of Anesthesiologists (ASA) I, II physical status

Exclusion Criteria:

* Patients' refusal.
* Critically ill patients.
* Patients who have contraindications to regional anesthesia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2020-10-24 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue score | 24 hours
  a scale to measure pain intensity graded from 0 = no pain to 10 = worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Esam A. Hamed, Asyut, Egypt